CLINICAL TRIAL: NCT06770179
Title: Effect of Ultrasound-assisted Lung Recruitment Maneuver on Preventing Perioperative Atelectasis, Prospective Randomized Study
Brief Title: Effect of Ultrasound-assisted Lung Recruitment Maneuver on Preventing Perioperative Atelectasis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Şeyma Karaduman Bulut, anesthetist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-83045809-604.01-904144
Record Dates: First submitted 2024-11-20; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Undergoing Surgery; Perioperatif Atelectasis
Keywords: perioperatif atelectasis; Recruitment maneuver; lung ultrasound

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1 (No Intervention): Patients in this group will receive a fixed PEEP of 5 cm H₂O during the perioperative period.
- group 2 (Experimental): In addition to the fixed PEEP of 5 cm H₂O, a recruitment maneuver will be performed at the end of the surgery.
  Interventions: Other: recruitment maneuver
- group 3 (Experimental): In addition to the fixed PEEP of 5 cm H₂O, a positional recruitment maneuver will be performed at the end of the surgery.
  Interventions: Other: positional recruitment maneuver

INTERVENTIONS:
Other: recruitment maneuver — in the group 2, in addition to the fixed PEEP of 5 cm H₂O, a recruitment maneuver is planned at the end of the surgery. This will involve administering 6 breaths with VC × 2, I/E ratio of 1:1, and a plateau pressure of less than 35 cm H₂O, before extubation.
  Arms: group 2
Other: positional recruitment maneuver — In the third group, in addition to the fixed PEEP, a recruitment maneuver will be performed at the end of the surgery before extubation. This will involve administering 6 breaths with VC × 2, I/E ratio of 1:1, and a plateau pressure of less than 35 cm H₂O, with 3 breaths in the right lateral decubitus position and 3 breaths in the left lateral decubitus position
  Arms: group 3

SUMMARY:
This study is based on the hypothesis that recruitment maneuver reduces perioperative atelectasis and associated complications, and lung ultrasonography can be used to detect this.

Patients aged 1 to 14 years with an ASA physical status classification of 1 to 3 and undergoing surgical procedures with a minimum duration of 2 hours will be included in the study.

Patients with an ASA physical status classification of 4, including those with defined pulmonary diseases (e.g., asthma requiring medication and having had two emergency visits in the past year), prematurity ( <36 weeks gestation / bronchopulmonary dysplasia), cystic fibrosis, diagnosed syndromic conditions, congenital cardiac diseases, abnormal chest X-rays, chest wall deformities, or a history of previous thoracic surgery, as well as those undergoing laparoscopic surgery, will be excluded from the study.

All patients will be premedicated with midazolam (0.05-1 mg/kg) if intravenous access is established, prior to transfer to the operating room. Upon arrival, standard monitoring will be initiated, including SpO2, ECG, and non-invasive blood pressure measurements. Following preoxygenation with 100% oxygen, induction will be performed using thiopental 5 mg/kg or propofol 2 mg/kg, fentanyl 2 mcg/kg, and rocuronium 0.6 mg/kg. After tracheal intubation, mechanical ventilation will be configured in pressure-controlled mode with a tidal volume of 8 ml/kg, PEEP of 5 cmH2O, FIO2 of 40%, and a respiratory rate adjusted to maintain ETCO2 within the range of 35-45 mmHg. Anesthesia maintenance will be achieved with sevoflurane and oxygen. During emergence, sugammadex 2 mg/kg will be administered as a neuromuscular reversal agent. The Aldrete scoring system will be employed for assessing patient readiness for transfer to the recovery unit.

GROUP 1: PEEP will be set at 5 cmH2O, and no recruitment maneuver will be performed.

GROUP 2: PEEP will be set at 5 cmH2O. Prior to extubation, a recruitment maneuver will be conducted with a Plato P max : 35 cmH2O, delivering 6 breaths at a vital capacity of 2 times, with an I/E ratio of 1:1.

GROUP 3: PEEP will be set at 5 cmH2O. Prior to extubation, a recruitment maneuver will be performed with a Plato P max : 35 cmH2O, delivering 3 breaths in the left lateral decubitus position and 3 breaths in the right lateral decubitus position, at a vital capacity of 2 times, with an I/E ratio of 1:1.

Lung ultrasonography will be performed at the following time points: 1) before induction, 2) at the 5-minute mark after induction, 3) before the recruitment maneuver, and 4) at the 5-minute mark after extubation.

The lungs will be assessed by dividing each hemithorax into 6 regions. Evaluation will include pleural sliding, A-lines, air bronchograms, B-score, and consolidation score. Both PLAPS points will be evaluated for B-score and consolidation score.

From the beginning of the operation, the following parameters will be recorded hourly: heart rate (HR), arterial blood pressure (ABP), oxygen saturation (SpO2), fraction of inspired oxygen (FIO2), end-tidal CO2 (ETCO2), peak pressure (Ppeak), PLATO pressure, delta pressure, and compliance.

During the postoperative 24-hour period, the following will be documented: temperature, desaturation, oxygen requirement, and the need for additional radiological investigations.

DETAILED DESCRIPTION:
Postoperative pulmonary complications are associated with increased mortality and morbidity. These complications occur in 2.8 % of all patients, and the rate can reach 14.5% in high-risk surgeries. Mechanical ventilation aims to improve gas exchange, reduce respiratory work, and provide sedation and muscle relaxation. While achieving these goals, it is crucial to avoid ventilator-induced lung injury. Given that approximately 234 million people are mechanically ventilated during anesthesia each year, reducing the effects of anesthesia and mechanical ventilation is of great importance. Therefore, efforts are ongoing to develop protective ventilation strategies during anesthesia.

The primary function of the lungs is to ensure adequate gas exchange by maintaining normal oxygen levels in the blood and eliminating carbon dioxide. This is achieved by optimizing lung volumes during the perioperative period. General anesthesia causes changes in respiratory physiology, affecting both oxygenation and carbon dioxide elimination. The effects of anesthesia on pulmonary function continue into the postoperative period, impacting pulmonary function. Factors influencing pulmonary function include loss of consciousness, ventilation mode, patient positioning, and the effects of anesthetic agents. These effects manifest as changes in lung volumes, airway resistance, and compliance, which in turn alter the ventilation/perfusion (V/Q) ratio. While newer agents used in anesthesia practice may have fewer side effects, they do not eliminate all the adverse effects of general anesthesia. A thorough understanding of pulmonary physiology helps in preventing potential complications during anesthesia and the postoperative period.

Atelectasis occurs in most patients under general anesthesia, with an incidence rate in children ranging from 68% to 100%. Respiratory complications, including atelectasis, are the most common adverse events in pediatric anesthesia. Smaller children and infants are particularly susceptible to hypoxemia due to their smaller residual capacities and increased metabolic demands. Atelectasis affects oxygenation in these children and exacerbates respiratory problems. This condition represents a significant issue that requires careful monitoring and intervention during surgery and anesthesia.

In recent years, lung ultrasound has been increasingly used for this purpose. It has a wide range of applications, including the verification of intubation, detection of pneumothorax, pleural effusion, pulmonary edema, and atelectasis.

Applying PEEP and performing recruitment maneuvers are beneficial for preventing atelectasis. However, data on the duration, frequency, and exact application of these techniques in pediatric age groups are limited.

Among the methods for detecting atelectasis, lung ultrasound is increasingly recognized as a rapid, simple, non-invasive, and radiation-free technique. Lung ultrasound has demonstrated reliable sensitivity and specificity in diagnosing anesthesia-related atelectasis in children .

The importance of preventing atelectasis, especially in the pediatric age group, is significant. Therefore, in our study, we aimed to assess the degree of anesthesia-related atelectasis in children using lung ultrasound and to evaluate the effectiveness of recruitment maneuvers in preventing respiratory complications

In the power analysis conducted before the study, based on previous studies, the minimum sample size required to achieve an effect size (f) of 0.4, a Type I error rate of 0.05, a Type II error rate of 0.20, and a power of 0.80 was found to be 66 participants. Considering a 20% dropout rate during the follow-up period, a total of 78 patients were decided to be included in the study.

Patients aged 1 to 14 years with an ASA physical status classification of 1 to 3 and undergoing surgical procedures with a minimum duration of 2 hours will be included in the study.

Patients with an ASA physical status classification of 4, including those with defined pulmonary diseases (e.g., asthma requiring medication and having had two emergency visits in the past year), prematurity ( < 36 weeks gestation / bronchopulmonary dysplasia), cystic fibrosis, diagnosed syndromic conditions, congenital cardiac diseases, abnormal chest X-rays, chest wall deformities, or a history of previous thoracic surgery, as well as those undergoing laparoscopic surgery, will be excluded from the study.

All patients will be premedicated with midazolam (0.05-1 mg/kg) if intravenous access is established, prior to transfer to the operating room. Upon arrival, standard monitoring will be initiated, including SpO2, ECG, and non-invasive blood pressure measurements. Following preoxygenation with 100% oxygen, induction will be performed using thiopental 5 mg/kg or propofol 2 mg/kg, fentanyl 2 mcg/kg, and rocuronium 0.6 mg/kg. After tracheal intubation, mechanical ventilation will be configured in pressure-controlled mode with a tidal volume of 8 ml/kg, PEEP of 5 cmH2O, FIO2 of 40%, and a respiratory rate adjusted to maintain EtCO2 within the range of 35-45 mmHg. Anesthesia maintenance will be achieved with sevoflurane and oxygen. During emergence, sugammadex 2 mg/kg will be administered as a neuromuscular reversal agent. The Aldrete scoring system will be employed for assessing patient readiness for transfer to the recovery unit.

GROUP 1: PEEP will be set at 5 cmH2O, and no recruitment maneuver will be performed.

GROUP 2: PEEP will be set at 5 cmH2O. Prior to extubation, a recruitment maneuver will be conducted with a Plato P max :35 cmH2O, delivering 6 breaths at a vital capacity of 2 times, with an I/E ratio of 1:1.

GROUP 3: PEEP will be set at 5 cmH2O. Prior to extubation, a recruitment maneuver will be performed with a Plato P max : 35 cmH2O, delivering 3 breaths in the left lateral decubitus position and 3 breaths in the right lateral decubitus position, at a vital capacity of 2 times, with an I/E ratio of 1:1.

Lung ultrasonography will be performed at the following time points: 1) before induction, 2) at the 5-minute mark after induction, 3) before the recruitment maneuver, and 4) at the 5-minute mark after extubation.

The lungs will be assessed by dividing each hemithorax into 6 regions. Evaluation will include pleural sliding, A-lines, air bronchograms, B-score, and consolidation score. Both PLAPS points will be evaluated for B-score and consolidation score.

From the beginning of the operation, the following parameters will be recorded hourly: heart rate (HR), arterial blood pressure (ABP), oxygen saturation (SpO2), fraction of inspired oxygen (FIO2), end-tidal CO2 (ETCO2), peak pressure (Ppeak), PLATO pressure, delta pressure, and compliance.

During the postoperative 24-hour period, the following will be documented: temperature, desaturation, oxygen requirement, and the need for additional radiological investigations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 to 14 years
* ASA scores of 1 to 3
* Minimum surgical duration of 2 hours.

Exclusion Criteria:

* Patients with an ASA score of 4,
* Defined lung diseases (such as those using medication for asthma and having a hospital visit within the past year)
* Prematurity ( bronchopulmonary dysplasia)
* Cystic fibrosis
* Diagnosed syndromic conditions
* Congenital cardiac disease
* Abnormal lung findings
* Chest wall deformities
* A history of chest surgery
* Those undergoing laparoscopic surgery

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
B scores | Perioperative (Lung ultrasound will be performed four times on each patient: T1: Pre-induction T2: 5 minutes after induction T3: Pre-recruitment maneuver T4: 5 minutes after extubation.)
  Each hemithorax will be divided into six regions using three longitudinal (parasternal, anterior axillary, and posterior axillary) and two transverse (1 cm above the nipple line and diaphragm) lines. Each region will be scanned sequentially from right to left, top to bottom, and front to back, with the probe perpendicular to the ribs. Pleural sliding, A-lines, air bronchograms, juxtapleural consolidation, and B-lines will be assessed. Additionally, B scores will be evaluated at two specific PLAPS points.
Consolidation Scores | Perioperative ( Lung ultrasound will be performed four times on each patient: T1: Pre-induction T2: 5 minutes after induction T3: Pre-recruitment maneuver T4: 5 minutes after extubation.)
  Each hemithorax will be divided into six regions using three longitudinal (parasternal, anterior axillary, and posterior axillary) and two transverse (1 cm above the nipple line and diaphragm) lines. Each region will be scanned sequentially from right to left, top to bottom, and front to back, with the probe perpendicular to the ribs. Consolidation scores will be evaluated at two specific PLAPS points

SECONDARY OUTCOMES:
HR | perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for HR will be recorded.
SpO₂ | perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for SpO₂ will be recorded.
MAP | Perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for MAP will be recorded.
ETCO2 | Perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for ETCO₂ will be recorded.
Peak P | Perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for Peak P will be recorded.
Plateau P | perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for Plateau P will be recorded.
Delta P | Perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values forDelta P will be recorded.
Compliance | perioperative
  Starting from the pre-induction period and continuing at 5 minutes after intubation and every subsequent hour, the values for compliance will be recorded.

OTHER OUTCOMES:
Postoperative Complications | Up to 24 Hours
  During the 24-hour postoperative period, fever, desaturation, oxygen requirements, and the need for additional radiological investigations will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi -Cerrahpaşa,Cerrahpaşa Tıp Fakültesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided